CLINICAL TRIAL: NCT01739127
Title: A Longitudinal Comparison of Aripiprazole vs. Higher Metabolic Risk Antipsychotic Drugs on Adiposity Using MRI
Brief Title: Comparison of Aripiprazole Versus Higher Metabolic Risk Antipsychotic Drugs on Adiposity Using MRI
Acronym: CALM
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: H12-01611
Record Dates: First submitted 2012-11-27; First posted 2012-12-03 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Psychotic Disorders; Bipolar Disorder; Metabolic Syndrome X
Keywords: Antipsychotic agents; Adverse effects; Magnetic Resonance Imaging
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Metabolic Syndrome | interventions — Aripiprazole; Risperidone; Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be offered the option of taking part in an optional biobanking component of the main study. Six milliliters of whole blood samples will be collected and stored at -80 degrees Celsius for genotyping to determine if certain genetic polymorphisms predispose individuals to gain weight while taking antipsychotic medications.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Aripiprazole: Participants receiving treatment with at least 10mg aripiprazole per day, as prescribed to them by their psychiatrists.
  Interventions: Drug: Aripiprazole
- Risperidone/Quetiapine: Participants receiving treatment with either risperidone or quetiapine, as prescribed to them by their psychiatrists.
  Interventions: Drug: Risperidone/Quetiapine
- Control: Healthy participants who are not taking any antipsychotic medications.

INTERVENTIONS:
Drug: Aripiprazole — To be prescribed and monitored by participant's attending physician (not given to participants as a part of the study).
  Other Names: ABILIFY
  Groups: Aripiprazole
Drug: Risperidone/Quetiapine — To be prescribed and monitored by participant's attending physician (not given to participants as a part of the study).
  Other Names: Risperdal; Apo-risperidone; Seroquel; Apo-quetiapine
  Groups: Risperidone/Quetiapine

SUMMARY:
The purpose of this study is to compare abdominal weight gain and fat distribution in people taking aripiprazole versus risperidone or quetiapine, to people not taking any of these antipsychotic medications.

DETAILED DESCRIPTION:
Second generation antipsychotic drugs have much greater efficacy for refractory schizophrenia and have much lower propensity to induce motor side-effects. These medications are seeing increased use for indications other than psychosis, and greater use in populations such as adolescents. However, one of the most critical issues in the field of psychiatry today is the overwhelming evidence that chronic use of the second generation antipsychotics can result in metabolic dysregulation, which includes weight gain, hyperlipidemia, and insulin resistance. A recent meta-analysis indicated that switching from other second generation antipsychotics to the antipsychotic drug aripiprazole consistently resulted in significant weight loss and may be an optimal treatment for patients who exhibit drug-induced weight gain. Therefore, we aim to compare metabolic dysregulation (namely abdominal weight gain and fat distribution)in participants taking aripiprazole, to participants who are taking higher-metabolic propensity antipsychotic drugs (such as risperidone or quetiapine), and to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 12+ years for healthy participants or participants with bipolar disorder; or aged 15+ years for participants with non-affective psychosis.
* Recent admission to hospital for psychiatric services related to first-episode psychosis or first-episode bipolar disorder.
* Participants being treated with an antipsychotic medication principally for psychosis or for bipolar disorder.
* Participants taking aripiprazole must be taking a dose of at least 10mg/day for the duration of the study.
* Participants must have received no more than 12 weeks of total lifetime exposure to antipsychotics.
* Participants may be in- or outpatients.
* Participants able to give informed consent, or informed consent through legally authorized representative.

Exclusion Criteria:

* Previous total lifetime exposure to antipsychotics of more than 12 weeks.
* Previously diagnosed with diabetes mellitus, seizure disorders, mental retardation (IQ < 70), or pregnancy (current or within 3 months postpartum).
* Participants who have been treated/are currently being treated with mood stabilizers (paroxetine, lithium, or valproic acid). Prior or concurrent use of Selective Serotonin Reuptake Inhibitor antidepressants (other than paroxetine) is acceptable.
* Received chemotherapy for cancer treatment in the 4 weeks prior to baseline or 16-week follow-up visit.
* Participants who are not able to fluently communicate in English.
* Contraindicated for MRI scan (i.e., has had major surgery in the last 6 months, morbid obesity, claustrophobia, and/or has metal in their bodies from a surgical intervention or working in metalwork, or is unsure if metal is present in their bodies, etc.).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have recently been seen at a community Early Psychosis Intervention (EPI) clinic, or at BC Children's Hospital for first-episode psychosis or bipolar disorder. Age-, sex-, and weight-matched controls will be recruited from the general community.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2012-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Abdominal distribution of visceral fat versus subcutaneous fat | Baseline (within 12 weeks of starting antipsychotic treatment), and 16 weeks later
  Change over time, and between groups, in amounts of visceral and subcutaneous fat as measured by automated segmentation of a magnetic resonance image (MRI).

SECONDARY OUTCOMES:
Fat content of the liver | Baseline (within 12 weeks of starting an antipsychotic), and 16 weeks later
  Change over time, and between groups, in the amount of fat accumulation in the liver as measured by magnetic resonance spectroscopy (MRS).
Metabolic measures | Baseline (within 12 weeks of starting an antipsychotic), and 16 weeks later
  Comparing change in the levels of hemoglobin, fasting lipid levels, adiponectin, leptin, insulin, and glucagon-like peptide 1 (GLP-1).
Glucose intolerance | Baseline (within 12 weeks of starting an antipsychotic), and 16 weeks later
  Change over time, and between groups, in ability to tolerate a glucose challenge as measured by an oral glucose tolerance test (OGTT).
Potential genetic factors of antipsychotic-induced weight gain | Sample to be taken after 16 weeks of participation in the study
  DNA will be extracted and amplified using polymerase chain reaction (PCR), and the presence or absence of certain single nucleotide polymorphisms will be identified by using primers.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair M Barr, Ph.D., Principal Investigator — The University of British Columbia
Locations (1):
- BC Mental Health & Addictions Research Institute, Vancouver, British Columbia, Canada